CLINICAL TRIAL: NCT03911531
Title: Whole Exome Sequencing and Whole Genome Sequencing for Nonimmune Fetal/Neonatal Hydrops
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Huda Al-Kouatly, Assistant Professor of Obstetrics and Gynecology, Thomas Jefferson University
Other Study IDs: IRB18D.728
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2024-11

CONDITIONS: Nonimmune Fetal Hydrops; Nonimmune Hydrops in Neonate; Genetic Disorders
Keywords: hydrops; prenatal diagnosis; amniocentesis; whole genome sequencing
MeSH Terms: conditions — Genetic Diseases, Inborn; Edema | interventions — Exome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from amniotic fluid samples and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fetuses: DNA obtained from amniotic fluid samples
  Interventions: Diagnostic Test: Whole Exome Sequencing; Diagnostic Test: Whole Genome Sequencing
- Neonates: DNA obtained from neonatal blood samples
  Interventions: Diagnostic Test: Whole Exome Sequencing; Diagnostic Test: Whole Genome Sequencing

INTERVENTIONS:
Diagnostic Test: Whole Exome Sequencing — Whole exome sequencing (WES) provides more detailed information through greater resolution, identifying single base-pair changes and small insertions and deletions. WES performs sequencing on the protein-coding exons, which are contained in 1-2% of the genome but make up over 85% of all known pathogenic mutations.
Diagnostic Test: Whole Genome Sequencing — Whole Genome Sequencing (WGS) has emerged in recent years as a diagnostic tool that sequences the entire genome and can pick up insertions or deletion of bases, structural variants and intronic single nucleotide variations.

SUMMARY:
Brief Summary: Nonimmune hydrops fetalis (NIHF) is a potentially fatal condition characterized by abnormal fluid accumulation in two or more fetal compartments. Numerous etiologies may lead to NIHF, and the underlying cause often remains unclear (1). The current standard of genetic diagnostic testing includes a fetal karyotype and chromosomal microarray (CMA), with an option to pursue single gene testing on amniocytes collected by amniocentesis (2). A large subgroup of the NIHF causes includes single gene disorders that are not diagnosed with the standard genetic workup for hydrops. Currently, nearly 1 in 5 cases of NIHF is defined as idiopathic, meaning there is no identified etiology (2). The investigators believe this is because the causes of NIHF are not completely investigated, specifically single gene disorders. Our research study aims to increase the diagnostic yield by performing whole exome sequencing (WES) and whole genome sequencing (WGS) on prenatal and neonatal NIHF cases when standard genetic testing is negative, identifying known and new genes, thus providing vital information to families regarding the specific diagnosis and risk to future pregnancies. The investigators plan to perform WES as the initial diagnostic test. If WES is negative, then the investigators will proceed to perform WGS.

DETAILED DESCRIPTION:
This is a prospective cohort study design for fetuses or neonates affected with NIHF. Mother-father-fetus trios of pregnancies complicated by idiopathic non-immune fetal hydrops will be identified. These patients will be counseled by a Maternal-Fetal Medicine specialist as would be the routine. As part of the routine work-up, amniocentesis will be recommended for karyotype, CMA and an infectious work-up. Amniocentesis will be performed by the Maternal-Fetal Medicine specialist of the referring institution. The patient will also be offered genetic counseling (routine). Subjects will be offered enrollment when inclusion criteria are met. After enrollment, the following samples will be collected: (1) maternal blood (2) paternal blood, (3) fetal DNA isolated from amniocytes (4) neonatal blood when referral is done postnatally. The WES results will be reported to the genetic counselor dedicated to the study. The parents will be contacted by the genetic counselor and counseled on the findings whether they were positive or negative. The result will also be communicated to the patient's primary MFM provider or pediatrician and appropriate referrals to pediatric genetics specialists will be made by the primary provider. In cases where no genetic disorder is identified, the sample will be stored and then subsequently whole genome sequencing will be performed.

ELIGIBILITY:
The following inclusion criteria will apply:

1. Fetal hydrops identified anytime in pregnancy after the first trimester
2. Parents are planning to proceed with amniocentesis as a routine workup for hydrops.
3. Both parents are available for blood sample collection
4. Normal CMA and normal karyotype if performed
5. Negative workup for Parvovirus B19, cytomegalovirus, toxoplasmosis, and syphilis
6. Negative fetomaternal hemorrhage workup as a cause for hydrops For cases of neonatal hydrops, the criteria for invasive prenatal testing will not be required as a postnatal blood sample from the hydropic infant will be the source of proband DNA.

The following exclusion criteria will apply:

1. Microarray was abnormal or karyotype was abnormal
2. Hydrops caused by congenital infection
3. Fetomaternal hemorrhage was a documented etiology for hydrops
4. Parental DNA cannot be obtained for either parents
5. Donor egg or donor sperm were utilized for conception
6. Fetus/Infant diagnosed with lysosomal storage disease
7. Pregnant woman or father of the baby less than 16 years of age
8. Hydrops was diagnosed concomitantly with intrauterine fetal demise

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from MFM physicians, paediatricians,and neonatologists.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify known single gene disorders that would not be detected by microarray as a cause of nonimmune fetal hydrops by performing whole exome sequencing (WES) | 5 years
Identify novel genetic disorders associated with nonimmune hydrops | 5 years

SECONDARY OUTCOMES:
Evaluate the incremental value of whole genome sequencing (WGS) in the evaluation of fetal hydrops when WES is negative | 5 years
Better counsel the parents about the etiology of hydrops especially if they desire a subsequent pregnancy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Huda B Al-Kouatly, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Society for Maternal-Fetal Medicine (SMFM); Norton ME, Chauhan SP, Dashe JS. Society for maternal-fetal medicine (SMFM) clinical guideline #7: nonimmune hydrops fetalis. Am J Obstet Gynecol. 2015 Feb;212(2):127-39. doi: 10.1016/j.ajog.2014.12.018. Epub 2014 Dec 31. PMID 25557883
- [Background] Whybra C, Mengel E, Russo A, Bahlmann F, Kampmann C, Beck M, Eich E, Mildenberger E. Lysosomal storage disorder in non-immunological hydrops fetalis (NIHF): more common than assumed? Report of four cases with transient NIHF and a review of the literature. Orphanet J Rare Dis. 2012 Nov 8;7:86. doi: 10.1186/1750-1172-7-86. PMID 23137060
- [Background] Lionel AC, Costain G, Monfared N, Walker S, Reuter MS, Hosseini SM, Thiruvahindrapuram B, Merico D, Jobling R, Nalpathamkalam T, Pellecchia G, Sung WWL, Wang Z, Bikangaga P, Boelman C, Carter MT, Cordeiro D, Cytrynbaum C, Dell SD, Dhir P, Dowling JJ, Heon E, Hewson S, Hiraki L, Inbar-Feigenberg M, Klatt R, Kronick J, Laxer RM, Licht C, MacDonald H, Mercimek-Andrews S, Mendoza-Londono R, Piscione T, Schneider R, Schulze A, Silverman E, Siriwardena K, Snead OC, Sondheimer N, Sutherland J, Vincent A, Wasserman JD, Weksberg R, Shuman C, Carew C, Szego MJ, Hayeems RZ, Basran R, Stavropoulos DJ, Ray PN, Bowdin S, Meyn MS, Cohn RD, Scherer SW, Marshall CR. Improved diagnostic yield compared with targeted gene sequencing panels suggests a role for whole-genome sequencing as a first-tier genetic test. Genet Med. 2018 Apr;20(4):435-443. doi: 10.1038/gim.2017.119. Epub 2017 Aug 3. PMID 28771251
- [Background] Taylor JC, Martin HC, Lise S, Broxholme J, Cazier JB, Rimmer A, Kanapin A, Lunter G, Fiddy S, Allan C, Aricescu AR, Attar M, Babbs C, Becq J, Beeson D, Bento C, Bignell P, Blair E, Buckle VJ, Bull K, Cais O, Cario H, Chapel H, Copley RR, Cornall R, Craft J, Dahan K, Davenport EE, Dendrou C, Devuyst O, Fenwick AL, Flint J, Fugger L, Gilbert RD, Goriely A, Green A, Greger IH, Grocock R, Gruszczyk AV, Hastings R, Hatton E, Higgs D, Hill A, Holmes C, Howard M, Hughes L, Humburg P, Johnson D, Karpe F, Kingsbury Z, Kini U, Knight JC, Krohn J, Lamble S, Langman C, Lonie L, Luck J, McCarthy D, McGowan SJ, McMullin MF, Miller KA, Murray L, Nemeth AH, Nesbit MA, Nutt D, Ormondroyd E, Oturai AB, Pagnamenta A, Patel SY, Percy M, Petousi N, Piazza P, Piret SE, Polanco-Echeverry G, Popitsch N, Powrie F, Pugh C, Quek L, Robbins PA, Robson K, Russo A, Sahgal N, van Schouwenburg PA, Schuh A, Silverman E, Simmons A, Sorensen PS, Sweeney E, Taylor J, Thakker RV, Tomlinson I, Trebes A, Twigg SR, Uhlig HH, Vyas P, Vyse T, Wall SA, Watkins H, Whyte MP, Witty L, Wright B, Yau C, Buck D, Humphray S, Ratcliffe PJ, Bell JI, Wilkie AO, Bentley D, Donnelly P, McVean G. Factors influencing success of clinical genome sequencing across a broad spectrum of disorders. Nat Genet. 2015 Jul;47(7):717-726. doi: 10.1038/ng.3304. Epub 2015 May 18. PMID 25985138
- [Derived] Rice SM, Varotsis DF, Wodoslawsky S, Critchlow E, Liu R, McLaren RA Jr, Makhamreh MM, Firman B, Berger SI, Al-Kouatly HB. Prenatal Phenotype of Alkuraya-Kucinskas Syndrome: A Novel Case and Systematic Literature Review. Prenat Diagn. 2024 Oct;44(11):1381-1397. doi: 10.1002/pd.6637. Epub 2024 Sep 3. PMID 39228063
- [Derived] Raymond M, Critchlow E, Rice SM, Wodoslawsky S, Berger SI, Hegde M, Empey PE, Al-Kouatly HB. Fetal pharmacogenomics: A promising addition to complex neonatal care. Mol Genet Metab. 2022 Sep-Oct;137(1-2):140-145. doi: 10.1016/j.ymgme.2022.08.002. Epub 2022 Aug 12. PMID 36029725